CLINICAL TRIAL: NCT04673292
Title: Community Collaboration to Combat COVID-19
Brief Title: Community Collaboration to Combat COVID-19 (C-FORWARD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00250298; P30AI094189-09S1 (NIH)
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Each household will be randomized to one of three arms in the study: Fixed site SOC testing (Arm 1), community-based, mobile van testing (Arm 2), or self-collected, home-based testing (Arm 3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed site SOC testing (Experimental): Fixed site Standard of Care (SOC) testing
  Interventions: Behavioral: Fixed site standard of care testing
- Community-based testing (Experimental): Community-based, mobile van testing
  Interventions: Behavioral: Community-based, mobile van testing
- Self-collected testing (Experimental): Self-collected, home-based testing
  Interventions: Behavioral: Self-collected, home-based testing

INTERVENTIONS:
Behavioral: Fixed site standard of care testing — This arm includes all three Johns Hopkins (JHMI) ambulatory outdoor testing sites across Baltimore City. Each site represents a traditional appointment-based scheduling system. Participants will be given a choice of 1 of 3 outdoor testing locations based on their preferences. Study staff will make an appointment for testing based on testing availability and participant schedule.
  Arms: Fixed site SOC testing
Behavioral: Community-based, mobile van testing — This arm offers the convenience of highly accessible testing and with the flexibility of no fixed appointment time. Each of the 12 geographic strata will have a single, centrally located testing site within the area, providing similar geographic access across households. The testing location will be published on the study website and social media so that participants can visit the location at a time convenient to them.
  Arms: Community-based testing
Behavioral: Self-collected, home-based testing — Individuals will receive a home-based testing kit delivered by a courier service as soon as the randomization of the household is complete. The kit will include provisions for contacting the courier service for pick up. Appropriate biohazard precautions are included. Each of the testing components of this kit will include FDA Emergency Use Authorization approved collection methods. Easy to use instructions with options to view pre-recorded videos and/or virtual 'on demand' coaching sessions with members of the study team via a HIPAA-secure Zoom session will be available.
  Arms: Self-collected testing

SUMMARY:
This is randomized trial where households will be randomized to identify the optimal SARS-CoV-2 (COVID-19) testing modality in a population-representative sample of households in Baltimore City, Maryland. 1,386 households in Baltimore City will be randomized 1:1:1 to one of three testing modalities: 1) fixed-site standard of care testing; 2) community-based mobile van testing; or 3) self-collected home, based testing.

DETAILED DESCRIPTION:
The target population will include English- and Spanish-speaking families residing in Baltimore City households (N=238,427). The sample size goal is 1,386 households (0.44% of households) or 3,000 individual household members. Households will be sampled using a multi-stage approach with 1) selection of 105 of 653 census block groups (CBGs) with probabilities proportional to the estimated number of occupied households selected from 9 strata of CBGs defined by socioeconomic status and race/ethnicity with over-sampling of CBGs with harder-to-reach populations (e.g., Latinos/x, low-income whites); 2) selection of residential addresses within each of the strata via non-linear optimization; and finally, 3) screening of individuals selected for eligibility (e.g., household occupied vs. not, English/Spanish speaking).

After completion of brief surveys, individuals will be asked to enroll other willing household members. One adult member of the household will be randomized 1:1:1 using a stratified, blocked approach with varying block sizes of 3, to one of three testing modalities: 1) fixed site standard of care testing; 2) community-based mobile van testing; or 3) self-collected home, based testing. Randomization will be stratified by geography (n=12 zones) and race/ethnicity (non-hispanic white/other, non-hispanic black and hispanic/latinx).

Arm 1 includes all three Johns Hopkins (JHMI) ambulatory outdoor testing sites across Baltimore City. Each site represents a traditional appointment-based scheduling system.

Arm 2 includes a convenient, accessible mobile van option which will be located in the center of each of 12 geographic zones.

Arm 3 includes a home-based testing kit which will be delivered by courier service.

Outcomes related to testing will be measured within 30 days of the initial randomization. Participants will be followed with weekly symptom pulses and monthly follow-up visits to ascertain subsequent testing need/COVID-19 symptoms. Testing during follow-up will be on-demand and participants can use either the fixed site or the home-based testing kits. The investigators will measure the impact of the time to receipt of SARS CoV-2 testing results.

ELIGIBILITY:
Inclusion Criteria for households

1. Selected address within Baltimore City
2. At least one member of the household >18 years of age who speaks English and/or Spanish
3. At least one member of the household provides informed consent
4. At least one member of the household psychologically fit to complete survey

Inclusion Criteria for Individuals

1. Reports primary residence within the sampled household
2. Provides informed consent
3. For children (12 years of age or older), with child assent.

Exclusion Criteria for households:

1. Adult member of the household is under the influence of illicit substances, in the opinion of the phone interviewer
2. Residents of nursing homes, half-ways houses or shelters
3. Psychologically unfit to complete the survey
4. Not a selected household address

Exclusion criteria for individuals

1. Person providing informed consent is under the influence of illicit substances

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Farley, PhD, MPH, NP, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- 2212 McElderry Street, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One person per household was enrolled
Units Other Than Participants: Households
Period: Overall Study
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing
Started | 277; 277 Households | 273; 273 Households | 281; 281 Households
Completed | 277; 277 Households | 273; 273 Households | 281; 281 Households
Not Completed | 0; 0 Households | 0; 0 Households | 0; 0 Households

BASELINE CHARACTERISTICS:
Units Other Than Participants: Households
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing | Total
Number analyzed (Participants) | 277 | 273 | 281 | 831
Number analyzed (Households) | 277 | 273 | 281 | 831
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [37 to 65] | 57 [39 to 67] | 56 [40 to 65] | 56 [39 to 65]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 199 | 182 | 192 | 573
  Male | 77 | 90 | 87 | 254
  Unknown | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 11 | 13 | 37
  Not Hispanic or Latino | 253 | 249 | 254 | 756
  Unknown or Not Reported | 11 | 13 | 14 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 6 | 5 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 118 | 122 | 119 | 359
  White | 137 | 132 | 143 | 412
  More than one race | 6 | 6 | 6 | 18
  Unknown or Not Reported | 5 | 7 | 8 | 20
Employment [Count of Participants; unit: Participants]
  Working now (either full or part time) | 162 | 144 | 151 | 457
  Retired/Disabled/Keeping House | 83 | 110 | 106 | 299
  Student | 6 | 5 | 5 | 16
  Unemployed | 19 | 9 | 19 | 47
  Other | 7 | 5 | 0 | 12
Essential Worker Status [Count of Participants; unit: Participants]
  Essential Worker | 67 | 64 | 63 | 194
  Not an Essential Worker | 195 | 201 | 209 | 605
  Unknown or Not Reported | 15 | 8 | 9 | 32
Educational Attainment [Count of Participants; unit: Participants]
  High School Graduate or Less | 60 | 69 | 63 | 192
  Some College Level/Technical/Vocational Degree/Associate's Degree | 62 | 60 | 66 | 188
  Bachelor's Degree | 45 | 62 | 54 | 161
  Other Advanced Degree | 109 | 80 | 96 | 285
  Unknown or Not Reported | 1 | 2 | 2 | 5
Health Insurance [Count of Participants; unit: Participants]
  No Health Insurance | 8 | 10 | 2 | 20
  Public (Medicare, Medicaid, Tricare) | 101 | 111 | 103 | 315
  Private (purchased directly or through employer) | 118 | 100 | 124 | 342
  Unknown or Not Reported | 50 | 52 | 52 | 154
History of COVID-19 Vaccination [Count of Participants; unit: Participants]
  Any COVID-19 Vaccination | 243 | 238 | 238 | 719
  No COVID-19 Vaccination | 31 | 33 | 41 | 105
  Unknown or Not Reported | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Uptake of SARS-CoV-2 Testing as Assessed by Proportion of Participants Who Complete Testing
Description: Uptake of SARS CoV-2 testing will be assessed by proportion of participants who are randomized and complete SARS CoV-2 testing.
Time Frame: Measured within 30 days of randomization/consent
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing
Number analyzed (Participants) | 277 | 273 | 281
Participants
  Completed PCR testing within 30 days of study randomization | 199 | 205 | 218
  Did not complete PCR testing within 30 days of randomization | 78 | 68 | 63
Statistical Analysis 1: Comparison: Fixed Site SOC Testing vs Community-based Testing; Test type: Equivalence — The fixed site SOC testing study arm was the standard of care and reference group. The null hypothesis was that there is not a statistically significant difference in the proportion of participants who complete PCR COVID-19 testing within 30 days of randomization when comparing community-based testing to the fixed site SOC testing; p = 0.67, Poisson Regression; Adjusted poisson regression was performed using Study Arm as a nominal variable in the model with the Fixed Site SOC Testing as the reference group; Prevalence Ratio = 1.04, 95% CI 2-sided [0.86 to 1.27]; Models were adjusted for employment
Statistical Analysis 2: Comparison: Fixed Site SOC Testing vs Self-collected Testing; Test type: Equivalence — The fixed site SOC testing study arm was the standard of care and reference group. The null hypothesis was that there is not a statistically significant difference in the proportion of participants who complete PCR COVID-19 testing within 30 days of randomization when comparing self-collected testing to the fixed site SOC testing; p = 0.43, Poisson Regression; [statistical method as in outcome 1, analysis 1]; Prevalence Ratio = 1.08, 95% CI 2-sided [0.89 to 1.31]; Models were adjusted for employment

2. Secondary Outcome: Time to Completion of SARS-CoV-2 Testing
Description: Time (In days) to completion of SARS CoV-2 testing from randomization
Time Frame: Measured from randomization to testing completion (within 30 days of randomization)].
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing
Number analyzed (Participants) | 277 | 273 | 281
days | 7 [5 to 11] | 6 [4 to 10] | 7 [5 to 12]
Statistical Analysis 1: Comparison: Fixed Site SOC Testing vs Community-based Testing; Times were censored at 30 days; Test type: Equivalence — Testing for equivalence in the difference in time from randomization to completion of SARS-CoV-2 PCR testing when comparing the community-based testing to fixed site SOC testing. Alpha threshold of 0.05; p = 0.14, Accelerated Failure Time — aprior significance threshold: p-value<0.05; Study Arm included as a nominal (dummy) variable in accelerated failure time models. Models adjusted for employment; Time Ratio = 0.87, 95% CI 2-sided [0.73 to 1.05]; Models adjusted for employment
Statistical Analysis 2: Comparison: Fixed Site SOC Testing vs Self-collected Testing; Times were censored at 30 days; Test type: Equivalence — Testing for equivalence in the difference in time from randomization to completion of SARS-CoV-2 PCR testing when comparing the self-collected testing arm to the fixed site SOC testing Alpha threshold of 0.05; p = 0.09, Accelerated Failure Time — aprior significance threshold: p-value<0.05; Study Arm included as a nominal (dummy) variable in accelerated failure time models. Models adjusted for employment; Time Ratio = 0.86, 95% CI 2-sided [0.71 to 1.03]; Models adjusted for employment

3. Secondary Outcome: Time From SARS CoV-2 Testing to Receipt of Results
Description: Time (in days) from SARS CoV-2 testing completion to the receipt of results by the participant.
Time Frame: Measured from testing completion to receipt of results (within 10 days of testing)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing
Number analyzed (Participants) | 277 | 273 | 281
days | 3 [1 to 6] | 3 [1 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Fixed Site SOC Testing vs Community-based Testing; Times were censored at 10 days; Test type: Equivalence — Null hypothesis: There is no significant difference in time from completion of SARS-CoV-2 test to receipt of SARS-CoV-2 test results when comparing the community-based testing to fixed site SOC testing; p = 0.56, Accelerated Failure Time — aprior threshold for significance: p<0.05; Study arm included as a nominal (dummy) variable in accelerated failure time models. Models adjusted for employment; Time Ratio = 0.96, 95% CI 2-sided [0.83 to 1.10]; Models adjusted for employment
Statistical Analysis 2: Comparison: Fixed Site SOC Testing vs Self-collected Testing; Times were censored at 10 days; Test type: Equivalence — Null hypothesis: There is no significant difference in time from completion of SARS-CoV-2 test to receipt of SARS-CoV-2 test results when comparing the self-collected testing arm to the fixed site SOC testing; p = 0.32, Accelerated Failure Time — aprior significance threshold: p-value<0.05; Study Arm included as a nominal (dummy) variable in accelerated failure time models. Models adjusted for employment; Time Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07]; Models adjusted for employment

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | Fixed Site SOC Testing | Community-based Testing | Self-collected Testing
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/273 | 0/281
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/273 | 0/281
Other Adverse Events (participants affected / at risk) | 0/277 | 0/273 | 0/281

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT04673292/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT04673292/ICF_001.pdf